CLINICAL TRIAL: NCT04277013
Title: Ultrasound Assessment of Gastric Content in Fasted Pregnant Women : a Prospective Study
Brief Title: Ultrasound Assessment of Gastric Content in Fasted Pregnant Women
Acronym: ECHOmater
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0560
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Gastric Ultrasound; Fasting ( 6H for Solid ; 2H for Clear Fluid ); Pregnant Women
Keywords: Anaesthesia; Obstetric; Diagnostic imaging; Stomach; Ultrasonography
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary aspiration of gastric content is one of the most feared perioperative complication of general anesthesia. Pregnant women are usually considered as high risk of pulmonary aspiration but there is no epidemiological study evaluating gastric content in pregnant women during the entire gestation periode.

The main objective is evaluating prevalency of "full stomach" in differents stages of pregnancy in fasted pregnant women.

DETAILED DESCRIPTION:
Subjects will be recruited at Montpellier University Hospital, from fasted pregnant women before surgery or from ultrasound exam performed during pregnancy.

ELIGIBILITY:
Inclusion criteria

An subject must fulfill all of the following criteria in order to be eligible for study enrollment:

* Aged at least 18 years old
* Pregnant women
* Fasted ( at least 6h for solid , 2h for clear fluid )

Exclusion criteria

* Previous Bariatric surgery / upper gastro-intestinal surgery
* Adult under protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Investigator would like to perform an ultrasound assessment of gastric content to every fasted pregnant women before surgery or during ultrasound exam happening during standard pregnancy monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative assessment of gastric content | 1 day
  Qualitative assessment of gastric content using "Perlas Grade

SECONDARY OUTCOMES:
Quantitative assessment of gastric content | 1 day
  Quantitative assessment of gastric content by measuring antral area
Feasibility evaluation of gastric ultrasound | pregnancy
  Feasibility evaluation of gastric ultrasound during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Christophe DADURE, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC